CLINICAL TRIAL: NCT00615732
Title: Prospective, Randomized Controlled Trial on the Effectiveness of Qigong and Exercise Therapy in Patients With Chronic Neck Pain
Brief Title: Qigong and Exercise for Neck Pain in Adults (QENA)
Acronym: QENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QENA-08
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Neck Pain
Keywords: qigong; traditional chinese medicine; exercise therapy; neck pain
MeSH Terms: conditions — Neck Pain | interventions — Qigong; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): qigong
  Interventions: Procedure: Qigong
- 2 (Active Comparator): exercise therapy
  Interventions: Procedure: exercise therapy
- 3 (No Intervention)

INTERVENTIONS:
Procedure: Qigong — 18 therapy sessions, during the first 3 months once a week, month 4 to 6 once every second week
  Arms: 1
Procedure: exercise therapy — 18 therapy sessions, during the first 3 months once a week, month 4 to 6 once every second week
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effectiveness of qigong for the treatment of chronic neck pain compared to exercise therapy and waiting list group.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic neck pain since at least 6 months and complaints for a maximum duration of 5 years
* neck pain more prominent than other pain in the spine
* average pain intensity of the last 7 days more or equal to 40 mm measured by a visual analogue scale (VAS 0 - 100 mm)
* normal mobility of the cervical spine
* intellectual and physical ability to participate in the study
* informed consent

Exclusion Criteria:

* cervical pain related to malignancy
* cervical pain due to an accident
* inflammatory joint disorders
* previous spine surgery
* protrusion/prolapse of a spinal disk, spondylolisthesis, with radicular symptomatology
* actually doing or planning to do other regular physical exercise during the study with possible positive effects on neck pain - such as swimming, yoga, pilates, tai chi, etc.
* use of pain drugs for other diseases (> 1x/week)
* pregnancy
* severe chronic or acute disease interfering with therapy attendance
* alcohol or substance abuse
* participation in another clinical trial in the last 6 months before study entry

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
average pain intensity during the last 7 days measured on a visual analogue scale (VAS) | baseline, 3, 6, 12, and 24 months

SECONDARY OUTCOMES:
Neck Pain and Disability Scale (NPAD, Wheeler 1999) | baseline, 3, 6, 12, and 24 months
health related quality of life (SF-36) | baseline, 3, 6, 12 and 24 months
patient expectation and self efficacy (questionnaire) | Baseline, 3, 6, 12, and 24 months
therapist's expectation | baseline, 3, 6, 12, and 24 months
undesired effects | 3, 6, 12, and 24 months
semi-structured interviews to detect changes due to therapy and to assess the used questionnaires | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany

REFERENCES:
- [Result] Rendant D, Pach D, Ludtke R, Reisshauer A, Mietzner A, Willich SN, Witt CM. Qigong versus exercise versus no therapy for patients with chronic neck pain: a randomized controlled trial. Spine (Phila Pa 1976). 2011 Mar 15;36(6):419-27. doi: 10.1097/BRS.0b013e3181d51fca. PMID 21178832